CLINICAL TRIAL: NCT04774042
Title: Probiotic Supplementation in the Dysbiosis of Bowel Preparation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202006016MIPB
Record Dates: First submitted 2021-02-19; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Microbial Colonization; Irritable Bowel Syndrome; Metabolic Syndrome
MeSH Terms: conditions — Communicable Diseases; Irritable Bowel Syndrome; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo HAC two packs once daily; Placebo Infloran one pill three times per day for 8 weeks
  Interventions: Dietary Supplement: Infloran placebo; Dietary Supplement: HAC placebo
- HAC (Experimental): Probiotic HAC two packs once daily; Placebo Infloran one pill three times per day for 8 weeks
  Interventions: Dietary Supplement: HAC probiotic; Dietary Supplement: Infloran placebo
- Infloran (Experimental): Placebo HAC two packs once daily; Probiotic Infloran one pill three times per day for 8 weeks
  Interventions: Dietary Supplement: Infloran probiotic; Dietary Supplement: HAC placebo

INTERVENTIONS:
Dietary Supplement: Infloran probiotic — Infloran
  Arms: Infloran
Dietary Supplement: HAC probiotic — HAc probiotic
  Arms: HAC
Dietary Supplement: Infloran placebo — Infloran placebo
  Arms: HAC; Placebo
Dietary Supplement: HAC placebo — HAC placebo
  Arms: Infloran; Placebo

SUMMARY:
Significant changes in gut microbiota was noted after the high-volume bowel preparation with PEG before colonoscopy. The dynamic changes were found to be short-term. However, the perturbation pattern of gut microbiota found after bowel preparation may link to metabolic syndrome and obesity. No study had investigated the supplementation of probiotic in this dynamic situation before. Here we proposed this study to fulfill the knowledge gap and also inquiry on the potential therapeutic strategy.1.To test the hypothesis of probiotic supplementation after bowel preparation alters the composition of gut microbiota in a short-term and long-term manner.2.To test the hypothesis of GI tract associated symptoms affected by probiotic supplementation after bowel preparation. 3. To test the hypothesis of clinical events, especially parameters of metabolic syndrome affected by probiotic supplementation after bowel preparation.

DETAILED DESCRIPTION:
Objectives: Colonoscopy is widely used for identification and treatment of colon polyps and intestinal symptoms. High-volume polyethylene glycol (PEG) bowel preparation prior to colonoscopy causes significant dysbiosis of gut microbiota. Currently dysbiosis of gut microbiota is associated with metabolic syndrome and obesity. However, inconclusive conclusions were drawn from clinical trials studying supplementary probiotics and beneficial clinical effects on metabolic parameters. However, no study has addressed the effects of probiotic supplementation on the labile and dynamic intestinal environment following bowel preparation. Aims: Our study aims at studying the short-term and long-term changes on gut microbiota following the probiotic supplementation after bowel preparation. We also aim at studying the changes in abdominal symptoms and parameters of metabolic syndrome. Methods: This study is a prospective, multicentered, randomized double blind three-armed placebo-controlled trial. Targeted population will be those undergoing PEG bowel preparation before colonoscopy. Each individual will be randomly assigned to one of the active probiotic or placebo supplementation. General health parameters and anthropometric measurements, stool, serum lab data, abdominal sonography, oral carnitine/choline challenge tests will be analyzed. The follow-up timepoints are pre- and post-bowel preparation, receiving probiotics/placebo for 8 weeks, 3 months and 6 months thereafter.Outcome measurement: Primary end point: Evaluate the chronological change of gut microbiota post-bowel preparation between probiotic group and placebo group. Secondary end points:To compare incidence of GI associated symptoms after taking probiotics between two groups. Also evaluate the effects of probiotic supplementation on parameters of metabolic syndrome, evaluate the effects on fatty liver and the interaction between SNP variation and the benefit of probiotic supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age >20
2. Undergoing colonofibroscopy (CFS) with PEG bowel preparation

Exclusion Criteria:

1. Inadequate bowel preparation
2. Subjects with active cancer or IBD (inflammatory bowel disease)
3. Subjects with history of abdominal surgery (including stomach, gallbladder, pancreas, small bowel, large bowel)
4. Subjects who take medication related to gastrointestinal motility within 1 months
5. Subjects who take antibiotics or probiotics within 1 months
6. Subjects under pregnancy
7. Allergic or intolerance to the study medication
8. Refused to randomization

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Alpha diversity | 32 weeks
  Change in alpha diversity of bacterial species post-bowel preparation between probiotic group and placebo group.
Beta diversity | 32 weeks
  Change in beta diversity of bacterial species post-bowel preparation between probiotic group and placebo group.
Bacterial species abundance | 32 weeks
  Change in abundance of bacterial species post-bowel preparation between probiotic group and placebo group.

SECONDARY OUTCOMES:
Incidence of functional bowel symptoms | 32 weeks
  Incidence of GI associated symptoms in 8 weeks (abdominal discomfort, diarrhea, constipation, bloating) after bowel preparation between probiotic group (L) and placebo group (P).
BMI | 32 weeks
  Change in BMI pre- and post-bowel preparation after probiotic or placebo supplementation
Insulin resistance | 32 weeks
  Change in HOMA-IR pre- and post-bowel preparation after probiotic or placebo supplementation
Dyslipidemia | 32 weeks
  Change in lipid profiles (T-CHO, LDL, HDL, TG in mg/dL) pre- and post-bowel preparation after probiotic or placebo supplementation
Total cholesterol | 32 weeks
  Change in Total cholesterol (mg/dL) pre- and post-bowel preparation after probiotic or placebo supplementation
LDL | 32 weeks
  Change in Low density lipoprotein, LDL (mg/dL) pre- and post-bowel preparation after probiotic or placebo supplementation
HDL | 32 weeks
  Change in high density lipoprotein, HDL (mg/dL) pre- and post-bowel preparation after probiotic or placebo supplementation
TG | 32 weeks
  Change in triglyceride, TG (mg/dL) pre- and post-bowel preparation after probiotic or placebo supplementation
Weight | 32 weeks
  Change in weight (Kg) pre- and post-bowel preparation after probiotic or placebo supplementation
Waist | 32 weeks
  Change in Waist (cm) pre- and post-bowel preparation after probiotic or placebo supplementation
Fatty liver (grade) | 32 weeks
  Change in fatty liver severity (grade) pre- and post-bowel preparation after probiotic or placebo supplementation
Fatty liver (CAP) | 32 weeks
  Change in fatty liver severity (CAP, dB/m) pre- and post-bowel preparation after probiotic or placebo supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Li-Chun Chang, M.D. Ph.D., Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No